CLINICAL TRIAL: NCT03732560
Title: A Retrospective Observational Study Comparing Nivolumab + Ipilimumab Combination vs. Nivolumab Monotherapy as First Line Treatment of Metastatic PD-L1 Positive Melanoma in the US
Brief Title: A Comparison of Nivolumab-based Treatments in a Real-world PD-L1 Positive Metastatic Melanoma Population in the US
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8RW
Record Dates: First submitted 2018-11-05; First posted 2018-11-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing treatment with nivolumab and ipilimumab
  Interventions: Other: Non-Interventional
- Patients undergoing treatment with nivolumab
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
The goal of this study is to describe patient characteristics, treatment outcomes and adverse events for patients with metastatic melanoma testing positive for PD-L1 expression treated first line (1L) with either nivolumab and ipilimumab in combination (NIVO + IPI) or nivolumab (NIVO) monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* First advanced of diagnosis of metastatic/Stage IV) melanoma
* Tested for PD-L1 expression with a tumor proportion score (TPS) greater than or equal to 1% (Phase 1 data collection)
* Initiating a first line of therapy during the index period between October 1, 2015 through July 1, 2017
* Medical history available for medical chart abstraction from date of diagnosis through most recent or current therapy (defined as end of data collection period)

Exclusion Criteria:

* Patients enrolled in a cancer treatment-related clinical trial prior to first line therapy initiation for metastatic/Stage IV) melanoma

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult metastatic melanoma patients with a positive PD-L1 expression level (above 1%) treated with nivolumab or nivolumab+ipilimumab in the first line setting in the US between Oct 1, 2015 and July 1, 2017
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) from Advanced Diagnosis | Minimum follow up 1 year

SECONDARY OUTCOMES:
Progression Free Survival (PFS) from Advanced Diagnosis | Minimum follow up 1 year
Overall Survival (OS) from 1L Therapy Initiation | Minimum follow up 1 year
Progression Free Survival (PFS) from Index Date | Minimum follow up 1 year
Objective Response Rate (ORR) | Minimum follow up 1 year
Best Therapy Response | Minimum follow up 1 year
  Best response (complete response, CR or partial response, PR) will be measured from the start of index treatment to progression or recurrence. Outcome will be reported as the percent of patients achieving best response from the total population of patients in a study arm.
Time to Best Therapy Response | Minimum follow up 1 year
Time to Loss of Peak Response | Minimum follow up 1 year
Response Evaluation Criteria in Solid Tumors (RECIST) | Minimum follow up 1 year
Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) criteria | Minimum follow up 1 year
Incidence of AE's | Minimum follow up 1 year
Incidence of SAE's | Minimum follow up 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Parsippany, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm